CLINICAL TRIAL: NCT02971124
Title: Observational Study to Assess Cognitive Performance in Elderly Life Via Meaning Play
Brief Title: Dr Solitaire: Assessing Cognitive Performance Through Meaningful Play
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S59650
Record Dates: First submitted 2016-11-09; First posted 2016-11-22 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: eHealth
Keywords: Cognitive Performance; Meaningful Play; Screening test; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Elderly
- Mild Cognitive Impaired Elderly

SUMMARY:
To assess cognitive performance by means of the game of Solitaire. In this study, the investigators want to define relevant game metrics, when playing Solitaire, that may be indicative of cognitive performance.

DETAILED DESCRIPTION:
12-15 healthy older persons will be observed, as well as 12-15 persons with cognitive impairment, while playing Solitaire. This will take the shape of contextual inquiries, i.e. the researcher visits the older person in his/her natural context and ask his/her to play Solitaire. Older persons will be observed playing 8-10 rounds of playing Solitaire, both with a physical deck of card and on a tablet. Gameplay actions and player behaviors will be observed and recorded for later analysis, via screen capturing software installed on the tablet, including the recordings of facial expressions and verbal utterances via the integrated touchpad camera and microphone. According to the contextual inquiry method, which is a 'light' form of participant observation, the researcher will take the role of an 'apprentice'; he/she will observe and may ask questions for a better understanding of the player actions. At the end of the visit, following cognitive domains will be measured through pen-and-paper testing: visual scanning and psychomotor speed (Digit symbol substitution test), attention and executive function (Trail making test, digit span, verbal fluency, maze test), Camden topographical memory,... The duration of such a visit will last approximately 120 minutes.

These observations of game play actions and behaviors and the results that participants obtained on the cognitive test battery will be analyzed with experts in light of cognitive performance. More particular, the investigator will look for the measurable aspects of cognitive performance in the game, guided by earlier measures put forward by Jimison et al and Kaye et al. While they still list generic measures (e.g. 'target detection' or 'correctly retrieving item from previous knowledge'), this study will now operationalize these specifically for the game of Solitaire and for the target group (e.g. 'detection of card to move onto the build stack' or 'retrieving the card as available from the pile'). Hence, possible game metrics will be discussed and defined.

ELIGIBILITY:
Inclusion Criteria:

For the HEALTHY participants

1. The participant has a minimum age of 65 years.
2. The participant is living independently or semi-independently at home, service flat or care home.
3. The participant has no subjective memory concern as reported by the participant, informant, or clinician.
4. The participant has a normal brain function documented by scoring above 27 on the MMSE, above 26 on the MOCA and has a score of 0 for the CDR.
5. In the opinion of the investigator, the participant is in stable medical condition and willing and able to perform study procedures in the opinion of the investigator.
6. The participant is fluent in written and verbal Dutch.

For the participants with COGNITIVE IMPAIRMENT:

1. The participant has a minimum age of 65 years.
2. The participant is living independently or semi-independently at home, service flat or care home.
3. In the opinion of the investigator, the participant is in stable medical condition and willing and able to perform study procedures in the opinion of the investigator.
4. The participant is fluent in written and verbal Dutch.
5. For MCI: MCI patients, at baseline, are diagnosed applying Petersen's diagnostic criteria, i.e., (1) cognitive complaint, preferably corroborated by an informant; (2) objective cognitive impairment, quantified as performance of more than 1.5 SD below the appropriate mean on the neuropsychological subtests (z-score below -1.5); (3) largely normal general cognitive functioning; (4) essentially intact activities of daily living (ADL) (basic and instrumental activities of daily living (iADL) were determined by a clinical interview with the patient and an informant); and (5) not demented.
6. For AD:Probable AD according to the National Institute on Aging/Alzheimer's Association Diagnostic Guidelines

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 24-30 participants, both cognitively healthy older persons (n = 12-15) as well as older persons with mild cognitive impairment (MCI) or mild Alzheimer's disease (mAD) (12-15)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Specification of Cognitive Performance Metrics for the game Solitaire | 1 day
  From this study, metrics will be defined which can measure cognitive performance in cardgames like Solitaire. Possible candidates are, but are not limited to: situational awareness to measure visual perception and performance on dual tasks to measure divided attention. A more detailed table of possible game metrics of cognitive performance can be found in H. B. Jimison, M. Pavel, P. Bissell, and J. McKanna, "A Framework for Cognitive Monitoring Using Computer Game Interactions," Medinfo 2007 Proc. 12th World Congr. Health Med. Inform. Build. Sustain. Health Syst., p. 1073, 2007.

SECONDARY OUTCOMES:
Design Guidelines Apps for the Elderly | 1 day
  While playing the Solitaire game, feedback considering the usability of the game can be used to formulate design guidelines for applications.

CONTACTS AND LOCATIONS:
Overall Officials: Vero Vanden Abeele, prof., Study Director — KU Leuven; Karsten Gielis, Drs., Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - Jessa Hospital, Hasselt, Limburg
  - University Hospital Leuven, Leuven, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gielis K, Vanden Abeele ME, De Croon R, Dierick P, Ferreira-Brito F, Van Assche L, Verbert K, Tournoy J, Vanden Abeele V. Dissecting Digital Card Games to Yield Digital Biomarkers for the Assessment of Mild Cognitive Impairment: Methodological Approach and Exploratory Study. JMIR Serious Games. 2021 Nov 4;9(4):e18359. doi: 10.2196/18359. PMID 34734825